CLINICAL TRIAL: NCT06828497
Title: Analgesic Efficacy of Quadratus Lumborum Block Against Erector Spinae Plane Block in Laparoscopic Sleeve Gastrectomy: a Prospective Randomized Study
Brief Title: Analgesic Efficacy of Quadratus Lumborum Block Against Erector Spinae Plane Block in Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Port Said University hospital (Other)
Responsible Party: Principal Investigator, Adel Ali Hassan, lecturer of anaesthesia and intensive cae, Port Said University hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT2023-014
Record Dates: First submitted 2025-02-11; First posted 2025-02-14 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Quadratus Lumborum Block; Erector Spinae Plane Block; Sleeve Gastrectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quadratus lumborum Block Group (Active Comparator): The patient was in the lateral position, and the US probe was placed in the anterior axillary line to visualize the typical triple abdominal layers. Then, the probe was placed in the midaxillary line, and at this juncture, the layers of abdominal layers started to taper. When the probe was placed in the posterior axillary line as per the posterior approach, sonoanatomy showed first the transversus abdominis disappearing, then the internal oblique and external oblique forming aponeurosis, and the appearance of the QL muscle was noticed. The posterior aspect of the QL muscle was confirmed, and a 22-G block needle was guided, in plane, and the needle tip was inserted into this aspect of the QL muscle. Following aspiration, the local anesthetic was injected into the lift behind the QL muscle. The same procedure was performed bilaterally
  Interventions: Procedure: Technique of erector spinae plane block:
- Erector spinae plane block Group (Active Comparator): The patient will be placed in a sitting position. Under aseptic conditions, a high-frequency linear transducer will be placed on the spinous process at the T8 level on the parasagittal plane and then slide 2.5-3 cm laterally to visualize the transverse process and erector spinae muscle. Using the in-plane technique, the needle was advanced between the transverse process and erector spinae muscle. The correct location was confirmed, and local anesthetic was injected between the muscle and transverse process. The same procedure was performed bilaterally
  Interventions: Procedure: Technique of posterior quadratus lumborum block (QL 2 block):

INTERVENTIONS:
Procedure: Technique of posterior quadratus lumborum block (QL 2 block): — The patient was in the lateral position, and the US probe was placed in the anterior axillary line to visualize the typical triple abdominal layers. Then, the probe was placed in the midaxillary line, and at this juncture, the layers of abdominal layers started to taper. When the probe was placed in the posterior axillary line as per the posterior approach, sonoanatomy showed first the transversus abdominis disappearing, then the internal oblique and external oblique forming aponeurosis, and the appearance of the QL muscle was noticed. The posterior aspect of the QL muscle was confirmed, and a 22-G block needle was guided, in plane, and the needle tip was inserted into this aspect of the QL muscle. Following aspiration, the local anesthetic was injected into the lift behind the QL muscle. The same procedure was performed bilaterally
  Arms: Erector spinae plane block Group
Procedure: Technique of erector spinae plane block: — The patient will be placed in a sitting position. Under aseptic conditions, a high-frequency linear transducer will be placed on the spinous process at the T8 level on the parasagittal plane and then slide 2.5-3 cm laterally to visualize the transverse process and erector spinae muscle. Using the in-plane technique, the needle was advanced between the transverse process and erector spinae muscle. The correct location was confirmed, and local anesthetic was injected between the muscle and transverse process. The same procedure was performed bilaterally
  Arms: Quadratus lumborum Block Group

SUMMARY:
The current investigation aimed to assess the postoperative analgesic efficacy of quadratus lumborum block against erector spinae plane block in sleeve gastrectomy surgeries

DETAILED DESCRIPTION:
In bariatric surgeries, overall pain is a conglomerate of three different and clinically separate components: incisional pain (somatic pain) due to trocar insertion sites, visceral pain (deep intra-abdominal pain), and shoulder pain due to peritoneal stretching and diaphragmatic irritation associated with carbon dioxide insufflation. Without effective treatment, this ongoing pain may delay recovery, mandate inpatient admission, and thereby increase the cost of such care.

The ultrasound-guided erector spinae plane (ESP) block influences both visceral and somatic pain; therefore, its use in laparoscopic surgeries and other abdominal surgeries can be advantageous. . ESP block is reported to lead to an analgesic effect on somatic and visceral pain by affecting the ventral rami and rami communicantes that include sympathetic nerve fibers, as local anesthetic spreads through the paravertebral space. When performed bilaterally, it can be as effective as thoracic epidural analgesia. Thoracic surgery and T seven level for abdominal surgeries. The number of surgeries involving multiple procedures and/or incisions is increasing, with such surgeries requiring complex analgesia protocols for pain management.

Currently, the Quadratus Lumborum (QL) block is performed as one of the perioperative pain management procedures for all generations (pediatrics, pregnant, and adult) undergoing abdominal surgery. The local anesthetic injected via the approach of the posterior QL block (QL 2 block) can more easily extend beyond the TAP to the thoracic paravertebral space or the thoracolumbar plane, producing somatic and visceral analgesia; the posterior QL block entails a broader sensory-level analgesic and may generate analgesia from T7 to L1

ELIGIBILITY:
Inclusion Criteria

* (ASA) I-III,
* age > 18 years and less than 60 years
* both sexes
* scheduled for laparoscopic sleeve gastrectomy under general anaesthesia

Exclusion Criteria:

* patient refusal,
* bleeding or coagulation abnormality
* local skin infection and sepsis at site of the block,
* hypersensitivity to the study drugs,
* body mass index > 50 kg/m²,
* Drug abuse, diabetes mellitus (DM), neurological or neuromuscular diseases, cardiovascular illnesses

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
the initial request for analgesia post-surgery | 24 hours
  analgesia request willbe assessed by Pain intensity was measured using the Visual Analogue Scale (VAS) score, the scale from 0 to 10 and 10 is the worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptian liver hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of the study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.